CLINICAL TRIAL: NCT05284747
Title: EVOLVE-MI: A Pragmatic Randomized Multicenter Trial of EVOLocumab Administered Very Early to Reduce the Risk of Cardiovascular Events in Patients Hospitalized With Acute Myocardial Infarction
Brief Title: EVOLVE-MI: EVOLocumab Very Early After Myocardial Infarction
Acronym: EVOLVE-MI
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Colorado Prevention Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190184; 2021-005272-19 (EudraCT Number)
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Cardiovascular Disease; Myocardial Infarction; Stroke; Coronary Revascularization
Keywords: Acute Myocardial Infarction; Cardiovascular Disease; Stroke; Coronary revascularization; Evolocumab; STEMI; NSTEMI; Heart Attack; Pragmatic
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Stroke; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction | interventions — evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Evolocumab + Routine Lipid Management (Experimental): Participants will receive open-label evolocumab every 2 weeks (Q2W) plus routine lipid management.
  Interventions: Drug: Evolocumab; Drug: Routine Lipid Management
- Routine Lipid Management (Active Comparator): Participants will receive routine lipid management per standard of care (SoC).
  Interventions: Drug: Routine Lipid Management

INTERVENTIONS:
Drug: Evolocumab — Evolocumab will be provided as a single-dose, prefilled autoinjector pen (AI/pen) for fixed dose subcutaneous (SC) injection.
  Other Names: Repatha; AMG 145
  Arms: Evolocumab + Routine Lipid Management
Drug: Routine Lipid Management — Routine lipid management therapies will be administered at the discretion of the investigator per SoC.

SUMMARY:
The primary objective of this study is to evaluate the effectiveness of early treatment with evolocumab plus routine lipid management vs routine lipid management alone when administered in the acute setting to reduce myocardial infarction, ischemic stroke, arterial revascularization, and all-cause death in subjects hospitalized for an acute myocardial infarction (non-ST-segment elevation myocardial infarction [NSTEMI] and ST-segment elevation myocardial infarction [STEMI]).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Hospitalized for primary reason of NSTEMI or STEMI due to presumed atherosclerotic disease

Exclusion Criteria:

* Participants requiring invasive hemodynamic and/or vasopressor/inotropic support at the time of screening
* Participants with elevated biomarkers of myocardial injury due to secondary/nonatherosclerotic etiology (eg, sepsis, atrial fibrillation, vasospasm, decompensated heart failure, uncontrolled hypertension, stress induced cardiomyopathy)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6019 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2027-05-29 (Estimated); Study Completion 2027-05-29 (Estimated)

PRIMARY OUTCOMES:
Total (first and subsequent) composite of myocardial infarction, ischemic stroke, any arterial revascularization procedure, and all-cause death | From Baseline to End of Study (Approximately 3.5 Years)

SECONDARY OUTCOMES:
Percentage Change From Baseline in LDL-C | From Baseline to Week 12
  Percent LDL-C change from baseline to 12 weeks in a subset of approximately 300 randomly selected participants.
Percentage Change From Baseline in LDL-C | From Baseline to Week 52
  Percent LDL-C change from baseline to 52 weeks in a subset of approximately 300 randomly selected participants.
Total (first and subsequent) composite of myocardial infarction, ischemic stroke, any arterial revascularization procedure, and cardiovascular death | From Baseline to End of Study (Approximately 3.5 Years)
Time to the First Occurrence of the Composite of Myocardial Infarction, Ischemic Stroke, any Arterial Revascularization Procedure, and All-Cause Death | From Baseline to End of Study (Approximately 3.5 Years)
Total Myocardial Infarctions Events | From Baseline to End of Study (Approximately 3.5 Years)
Total Arterial Revascularization Procedures | From Baseline to End of Study (Approximately 3.5 Years)
Total Ischemia-driven Coronary Revascularization Procedures | From Baseline to End of Study (Approximately 3.5 Years)
Total Ischemic Strokes | From Baseline to End of Study (Approximately 3.5 Years)
Time to Cardiovascular Death | From Baseline to End of Study (Approximately 3.5 Years)
Time to All-Cause Death | From Baseline to End of Study (Approximately 3.5 Years)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (120):
- United States (81):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Eastern Shore Research Institute, Fairhope, Alabama
  - Heart Center Research LLC, Huntsville, Alabama
  - Northern Arizona Healthcare Corporation Cardiovascular Institute, Flagstaff, Arizona
  - Scottsdale Healthcare at Shea - HonorHealth, Scottsdale, Arizona
  - Pima Heart and Vascular Clinical Research, Tucson, Arizona
  - John Muir Health and Cardiovascular Institute, Concord, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - University of California-Irvine, Orange, California
  - University of Colorado Hospital, Aurora, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Cardiology Associates of Fairfield County PC, Stamford, Connecticut
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - University of Florida at Gainesville, Gainesville, Florida
  - University of Florida and Shands Hospital, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Cardiology Partners Clinical Research Institute, Palm Beach Gardens, Florida
  - Baptist Health Care, Pensacola, Florida
  - Ascension Sacred Heart, Pensacola, Florida
  - Clearwater Cardiovascular Consultants, Safety Harbor, Florida
  - Tampa Cardiovascular Interventions and Research, Tampa, Florida
  - Clinical Site Partners Orlando dba Flourish Research, Winter Park, Florida
  - Saint Lukes Boise Medical Center, Boise, Idaho
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Ascension Saint Vincent Heart Center, Indianapolis, Indiana
  - Reid Physician Associates, Richmond, Indiana
  - University of Kansas Hospital, Kansas City, Kansas
  - Midwest Heart and Vascular Specialists, Overland Park, Kansas
  - University of Louisville Health - Jewish Hospital, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Healthy Heart Cardiology, Grand Rapids, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - McLaren Macomb Research Services, Mount Clemens, Michigan
  - McLaren Northern Michigan Hospital, Petoskey, Michigan
  - Advanced Cardiology Associates, Rochester Hills, Michigan
  - Essentia Health Saint Marys Medical Center, Duluth, Minnesota
  - Jackson Heart, Jackson, Mississippi
  - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - Saint Lukes Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, North Kansas City, Missouri
  - Advanced Heart Care LLC, Bridgewater, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Michaels Medical Center, Newark, New Jersey
  - South Shore University Hospital Northwell Health, Bay Shore, New York
  - New York Presbyterian-Weill Cornell Medical Center, New York, New York
  - Hudson Valley Cardiovascular Practice PC, Poughkeepsie, New York
  - University of Rochester Medical Center, Rochester, New York
  - Richmond University Medical Center, Staten Island, New York
  - Stony Brook Medicine, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina Cardiology, Chapel Hill, North Carolina
  - Novant Health Heart and Vascular Institute Presbyterian Medical Center, Charlotte, North Carolina
  - Moses H Cone Memorial Hospital, Greensboro, North Carolina
  - Aultman Hospital, Canton, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Genesis Healthcare System, Zanesville, Ohio
  - Ascension Saint John Bartlesville, Tulsa, Oklahoma
  - Ascension Saint John Tulsa, Tulsa, Oklahoma
  - Wellspan Chambersburg Hospital, Chambersburg, Pennsylvania
  - Lancaster General Hospital/The Heart Group of Lancaster, Lancaster, Pennsylvania
  - Reading Hospital Tower Health, West Reading, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Kent Hospital, Warwick, Rhode Island
  - Prisma Upstate and Midlands Greenville Hospital System, Columbia, South Carolina
  - Upstate Cardiology, Greenville, South Carolina
  - Tennova Healthcare-Turkey Creek Medical Center, Knoxville, Tennessee
  - Ascension Saint Thomas Nashville, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Parkway Cardiology Associates, Oak Ridge, Tennessee
  - Cardiovascular Research of Knoxville North Knoxville Medical Center, Powell, Tennessee
  - Ascension Texas Cardiovascular, Austin, Texas
  - Ascension Texas Cardiovascular Kyle, Kyle, Texas
  - Bon Secours St Marys Hospital Richmond, Midlothian, Virginia
  - Chippenham Hospital, Richmond, Virginia
  - Aurora Saint Lukes Medical Center, Milwaukee, Wisconsin
- Brazil (24):
  - Clínica Silvestre Sante, Rio Branco, Acre
  - Instituto Cardiovascular de Linhares, Linhares, Espírito Santo
  - Hospital Ruy Azeredo, Ipiranga Goiânia, Goiás
  - Hospital Universitario Sao Francisco na Providencia de Deus, Ipiranga Goiânia, Goiás
  - Hospital Madre Teresa, Belo Horizonte, Minas Gerais
  - Hospital Universitário Ciências Médicas de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Hospital do Coracao de Pocos de Caldas CEC servicos medicos, Poços de Caldas, Minas Gerais
  - Ps Cardiologico de PE - Procape, Casa Forte, Pernambuco
  - Instituto Atena de Pesquisa Clínica, Natal, Rio Grande do Norte
  - Centro de Pesquisa Clínica Associação Hospitalar Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Santa Casa de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Mãe de Deus, Porto Alegre, Rio Grande do Sul
  - Hospital Beneficência Portuguesa, São Paulo, Rio Grande do Sul
  - Cmep-Centro Multidisciplinar Ensino e Pesq, Joinville, Santa Catarina
  - Instituto de Cardiologia de Santa Catarina, Praia Comprida, Sao Jose, Santa Catarina
  - Centro de Pesquisa Clinica do Coracao, Aracaju, Sergipe
  - Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - Irmandade da Santa Casa de Misericordia de Marilia, Marília, São Paulo
  - Hospital Regional de Presidente Prudente, Presidente Prudente, São Paulo
  - Instituto Dante Pazanesse, São Paulo, São Paulo
  - Instituto do coracao da Faculdade de Medicina da Universidade de Sao Paulo - InCor, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
- Sweden (15):
  - Alingsas Lasarett, Alingsås
  - Gavle Sjukhus, Gävle
  - Lanssjukhuset Ryhov, Jönköping
  - Blekingesjukhuset Karlskrona, Karlskrona
  - Linkoping University Hospital, Linköping
  - Sunderby Sjukhus, Luleå
  - Skane Universitetssjukhus i Lund, Lund
  - Molndals Sjukhus, Molndahl
  - Vrinnevisjukhuset, Norrkoeping, Norrköping
  - Ostersunds sjukhus, Östersund
  - Sodersjukhuset, Stockholm
  - Sundsvalls Sjukhus, Sundsvall
  - Akademiska Sjukhuset i Uppsala, Uppsala
  - Centrallasarettet Vaxjo, Vaxjo
  - Vastmanlands Sjukhus Vasteras, Västerås

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com